CLINICAL TRIAL: NCT06733155
Title: Pragmatic Randomized Trial to Evaluate the Impact of Various Interventions to Increase the Uptake of Surveillance Mammography in Eligible Women in Singapore
Brief Title: Trial to Evaluate the Impact of Various Interventions to Increase the Uptake of Surveillance Mammography in Eligible Women in Singapore
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023/01007
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2024-10

CONDITIONS: This Study Evaluates Interventions to Increase Surveillance Mammography Uptake for Early Breast Cancer Detection Among Singaporean Women
Keywords: Breast Neoplasms; Mammography
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This study follows a parallel assignment model where participants are randomly assigned to one of five distinct arms: a control arm or one of four intervention arms. Each arm receives a different intervention, and the effects are compared to assess the impact on the uptake of surveillance mammography.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Observational Arm (No Intervention): Does not receive any mailer reminder to go for mammogram.
- Arm 1 (control) (Experimental): Receives a mail reminder with basic information about breast cancer and instructions on scheduling a mammogram
  Interventions: Other: Only reminder mailer
- Arm 2: Financial incentive (Experimental): Receives mail reminder + a $10 voucher for completing a mammogram within three months.
  Interventions: Other: Financial intervention
- Arm 3: Lottery incentive (Experimental): Receives mail reminder + chance to win a $5000 lottery for completing the screening within three months.
  Interventions: Other: Lottery intervention
- Arm 4: Health messaging (Experimental): Receives mail reminder + QR code to a 60-second video from an influential person, available in four languages (English, Chinese, Malay, Tamil).
  Interventions: Other: Health Messages
- Arm 5: Personal Health Concierge (Experimental): Receives mail reminder + a dedicated hotline for scheduling mammograms with the help of a health concierge over eight weeks.
  Interventions: Other: Personal Health Concierge

INTERVENTIONS:
Other: Financial intervention — Participants completing the mammogram within the study end date will receive a $10 voucher.
  Arms: Arm 2: Financial incentive
Other: Lottery intervention — Participants completing the mammogram within the study end date will receive achance to win a $5000 lottery.
  Arms: Arm 3: Lottery incentive
Other: Health Messages — Participants will receive a less than 5 minute long video from an influential person. The video will be available in four languages (English, Chinese, Malay, Tamil).
  Arms: Arm 4: Health messaging
Other: Personal Health Concierge — Participants will be able to call a dedicated hotline for scheduling mammograms with the help of a health concierge over eight weeks of receive the the mailer.
  Arms: Arm 5: Personal Health Concierge
Other: Only reminder mailer — Receives a mail reminder with basic information about breast cancer and instructions on scheduling a mammogram.
  Arms: Arm 1 (control)

SUMMARY:
Breast cancer is the most common cancer among women in Singapore, with more than 70 women out of every 100,000 being diagnosed each year. Early detection through regular mammograms can significantly reduce deaths from breast cancer. Although Singapore has had a national breast cancer screening program (now part of the Screen for Life initiative) for over 20 years, and the government offers substantial subsidies to make screening more affordable, participation remains low at only 30-40%. This low uptake is due to factors like fear, lack of awareness, cultural beliefs, and a perceived low risk of breast cancer. To be effective on a large scale, at least 70% of women need to participate in regular mammography screenings. While researchers in Singapore and Asia have studied the reasons behind low screening rates, there is still a lack of large-scale studies that test different strategies to increase mammography participation in these regions.

This trial will recruit 12,000 women aged 50-69 who have not undergone a mammogram in the past two years. 9000 women will be randomized into five intervention arms. The interventions include: direct mail reminder (Arm 1, control, n=3000), financial incentive (Arm 2, n=1500), lottery incentive (Arm 3, n=1500), health messaging from an influential figure (Arm 4, n=1500), and personal health concierge for appointment scheduling (Arm 5, n=1500). Another 3000 women will be placed in a non-interventional arm (NI arm) for observational analysis, that receives no reminders at all. A post-intervention telephone survey will assess intervention effectiveness.

The primary outcome is mammogram uptake across intervention arms with Arm 1 as a reference. Secondary outcome will be to compare Arm 1 with NI arm. Subgroup analyses will evaluate differences in uptake by sociodemographic factors, such as ethnicity and socioeconomic status. A cost-effectiveness analysis will assess the financial viability of each intervention.

This is the first large-scale study in Singapore and Asia to compare multiple interventions to boost mammography uptake. Findings will provide evidence-based strategies to improve breast cancer screening participation, potentially reducing breast cancer mortality and informing future public health policy.

DETAILED DESCRIPTION:
This study aims to evaluate different interventions to boost breast cancer screening (mammography) participation among women in Singapore, aged 50-69, using data from the National University Health System (NUHS). 9000 eligible women will be randomized into one control arm and four experimental arms, receiving different combinations of reminders and incentives. Another 3000 women will be placed in an observational arm that receives no reminders at all. The study will use data from the NUHS electronic health records (EPIC) and NUHS app to monitor mammogram completion rates, exploring the effectiveness of each intervention.

Study Arms:

Control Group (Direct Mail Reminder): Receives a mail reminder with basic information about breast cancer and instructions on scheduling a mammogram.

Financial Incentive Group: Mail reminder + a $10 voucher for completing a mammogram within three months.

Lottery Incentive Group: Mail reminder + chance to win a $5000 lottery for completing the screening within three months.

Health Messaging Group: Mail reminder + QR code to a 60-second video from an influential person, available in four languages (English, Chinese, Malay, Tamil).

Personal Health Concierge Group: Mail reminder + a dedicated hotline for scheduling mammogram with the help of a health concierge over eight weeks.

Selection and Randomization:

Eligible participants will be selected from over 500,000 registered users of the OneNUHS app. Randomization will be done using a random number generator, with control and experimental arms receiving a 2:1 ratio. Data collected include basic demographic details and mammogram history, extracted securely from the EPIC system.

Data Collection:

Women in each arm will receive a physical mailer and three push notifications over three weeks, instructing them to schedule a mammogram at any approved screening center. Data on mammogram attendance will be extracted from EPIC post-study, and a subset of participants will be surveyed to gather feedback.

Primary and Secondary Endpoints:

The study will compare mammogram participation rates between the control and experimental arms, with secondary analyses exploring the uptake rates of arm 1 and NI arm as well as, impact of ethnicity, age, and income (via housing type) on outcomes. Additionally, a cost-effectiveness analysis will assess the impact of interventions on breast cancer detection and healthcare savings.

Follow-up and Evaluation:

A post-trial telephone survey of 750 participants will gather insights into their response to the interventions. The study aims to provide actionable insights into effective, scalable interventions to improve mammography uptake and reduce breast cancer mortality in Singapore.

ELIGIBILITY:
Inclusion Criteria:

* Singaporean citizen
* Age 50-69
* Registered as a patient at the National University Hospital
* Registered and active user of OneNUHS App
* Signed up with Healthier SG with a primary care provider within the NUHS Primary Care Network

Exclusion Criteria:

* Diagnosis of breast cancer in EPIC
* Mammogram done in the past 24 months in EPIC

Ages: 50 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12000 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of Mammogram Uptake Between Intervention Arms (2-5) and Control Arm | 3 month from study start or 4 months from randomization
  Primary endpoint: Comparison of the proportion of women who undergo surveillance mammography among participants in Arms 2-5 versus Arm 1 (control arm).

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee SC, Lucky SS, Zhu J, Ow S, Loh L, Tan JH, Lim SE, Hairom Z, Mehta S, Tai BC, Goh BC. Pragmatic Interventions to Boost Surveillance Mammogram Uptake Among an Overdue Population: A Randomized Clinical Trial. JAMA Intern Med. 2026 Jan 1;186(1):27-35. doi: 10.1001/jamainternmed.2025.5873. PMID 41212556